CLINICAL TRIAL: NCT04629651
Title: Phase I/II Prospective Trial Investigating the Safety and Efficacy of Captopril Use on the Degree of Marrow Fibrosis in Patients With Primary or Secondary Bone Marrow Fibrosis/Myeloproliferative Neoplasms
Brief Title: Captopril Use on the Degree of Marrow Fibrosis in Bone Marrow Fibrosis/Myeloproliferative Neoplasms
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI discretion
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3920
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Bone Marrow Fibrosis; Myeloproliferative Neoplasm
Keywords: primary myelofibrosis (PMF); post-polycythemia vera/essential thrombocythemia-MF (secondary MF)
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — Captopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Captopril (Experimental): In phase I, Cohorts of 3 patients each will receive doses of captopril with a goal dose of 150mg total by mouth (PO) daily. Initial dose per patient will start at 12.5 mg daily, which will then be increased on weekly intervals as tolerated. To be administered per the intra-patient dose escalation scheme below
  Phase I:
  Day 0: 12.5mg/day Day 7: 12.5mg twice daily Day 14: 12.5mg three times daily Day 21: 25mg three times daily Day 28: 50mg three times daily
  Phase II: The efficacy of captopril will be assessed in the Phase II portion. Captopril given at Maximum Tolerated Dose - bone marrow evaluation to be done at 6 months
  Interventions: Drug: Captopril

INTERVENTIONS:
Drug: Captopril — Oral, to be administered per the dose escalation scheme.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of captopril and evaluate the effectiveness captopril as measured by changes in the grade of bone marrow scar tissue. The change in spleen size by ultrasound will also be measured.

DETAILED DESCRIPTION:
Captopril is an investigational (experimental) drug that works by inhibiting the production of angiotensin II by blocking angiotensin converting enzyme. Reducing angiotensin II may reduce the bone marrow scar tissue in myelofibrosis. It is not approved by the Food and Drug Administration (FDA) for this indication. Participants in this study will be asked to have 2 bone marrow biopsies, a total of 3 blood samples, and fill out questionnaires asking about how you feel.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed diagnosis of primary myelofibrosis (PMF), or post-polycythemia vera/essential thrombocythemia-MF (i.e. secondary MF) by 2016 WHO criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 -2
* Creatinine clearance >30 ml/minute
* Women of childbearing potential should be advised to avoid becoming pregnant while receiving treatment. All men and women of childbearing potential must use acceptable methods of birth control throughout the study.
* Participants should be able to give voluntary informed written consent to participate in the study. Informed consent will be obtained prior to enrollment and before any study-related procedure is done that is not part of standard medical care, with the understanding that consent may be withdrawn by the participants any time without prejudice to future medical care.

Exclusion Criteria:

* Completed hematopoietic cell transplant (HCT)
* Presence of >10% blasts in peripheral blood or on bone marrow examination
* Screening blood pressure(BP)parameters of systolic BP < 100 and diastolic BP < 60
* Splenic irradiation within 3 months prior to the first dose of captopril
* Prior ACE inhibitor, angiotensin II receptor antagonist, or aliskiren use within 12 months prior to trial enrolment
* Known allergy/hypersensitivity to ACE inhibitors
* Participants receiving any other investigational agents
* Pregnant or nursing participants - captopril is a risk category D and is excreted in breast milk
* Participants with creatinine clearance <30 ml/minute or on dialysis
* Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in degree of bone marrow fibrosis by World Health Organization WHO grade | At 6 months
  Change in degree of bone marrow fibrosis by WHO grade. "Change" is defined as reduction by one grade (e.g. MF-3 to MF-2 or MF-2 to MF-1)

SECONDARY OUTCOMES:
Change in spleen size by ultrasound | At 3 months
  Change in spleen size in centimeters measured using abdominal ultrasound by an experienced radiologist. Spleen length will be asses for response
Change in spleen size by ultrasound | At 6 months
  Change in spleen size in centimeters measured using abdominal ultrasound by an experienced radiologist. Spleen length will be asses for response
Change in symptom burden assessed using Myeloproliferative Neoplasm Symptom Assessment Form total symptom scores (MPN-SAF TSS) | At 3 months
  Change in symptom burden assessed using MPN-SAF TSS The MPN-SAF TSS is assessed by the patients themselves and this includes fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers. Scoring is from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be) for each item. The MPN-SAF TSS is the summation of all the individual scores (0-100 scale). Symptoms response requires ≥50% reduction in the MPN-SAF TSS.
Change in symptom burden assessed using MPN-SAF TSS | At 6 months
  Change in symptom burden assessed using Myeloproliferative Neoplasm Symptom Assessment Form total symptom scores (MPN-SAF TSS).
  The MPN-SAF TSS is assessed by the patients themselves and this includes fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers. Scoring is from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be) for each item. The MPN-SAF TSS is the summation of all the individual scores (0-100 scale). Symptoms response requires ≥50% reduction in the MPN-SAF TSS.
Response rate per International Working Group-Myeloproliferative Neoplasms Research and Treatment 2 (IWG-MRT) Criteria as measured by percent of participants with CR, PR, or CI | Up to 1 year from end of treatment
  Includes Complete response (CR), partial remission (PR) or Clinical improvement (CI)
  CR: Bone marrow: Age-adjusted normocellularity; <5% blasts; ≤grade 1 MF
  AND
  Peripheral blood: Hemoglobin ≥10 g/dL and <upper normal limit (UNL); Neutrophil count ≥1 x 10^9/L and <UNL; Platelet count ≥100 x 10^9/L and <UNL;<2% immature myeloid cells Clinical: Resolution of disease symptoms; Spleen & liver not palpable; No evidence of extramedullary hematopoiesis (EMH)
  PR: Periph. blood: Hem. ≥10 g/dL and <UNL; Neutrophil count ≥1 x 10^9/L and <UNL; Platelet count ≥100 x 10^9/L & <UNL;<2% immature myeloid cells
  OR
  Bone marrow: [See CR]
  AND
  Peripheral blood: Hem. ≥85, but <10 g/dL & <UNL; Neutrophil count ≥1 x 10^9/L & <UNL; Platelet count ≥50, but <100 x 109/L and <UNL; <2% immature myeloid cells Clinical:[See CR]
  CI: Achievement of anemia, spleen, or symptoms response without progressive disease or increase in severity of anemia, thrombocytopenia, or neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Gerds, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make all individual participant data (IPD) and related data dictionaries available. We will also make the protocol available.
Supporting Information: Study Protocol